CLINICAL TRIAL: NCT05634941
Title: Effect of Transcranial Direct Current Stimulation of the Greater Occipital Nerve on Memory Function Improvement and and the Locus Coeruleus-Noradrenergic Circuits in Stable Depression Patients
Brief Title: Effect of ON-tDCS on Memory Function Improvement and Related Circuits in Stable Depression Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT20221169
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Depression
Keywords: Depression; transcranial direct current stimulation; the locus coeruleus-noradrenergic circuit
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active ON-tDCS (Active Comparator): The active group will receive the active transcranial direct current stimulation via a saline-soaked pair of surface sponges. Patients received this treatment protocol for 5 consecutive days.
  Interventions: Device: Active ON-tDCS
- Sham ON-tDCS (Sham Comparator): The sham group will also receive the transcranial direct current stimulation for 5 consecutive days on sham procedure. The rationale behind this sham procedure was to mimic the transient skin sensation at the beginning of active ON-tDCS without producing any conditioning effects on the brain.
  Interventions: Device: Sham ON-tDCS

INTERVENTIONS:
Device: Active ON-tDCS — DC was transmitted via a saline-soaked pair of surface sponges and delivered by specially developed, battery-driven, constant current stimulator with a maximum output of 2 mA. For each participant receiving ON-tDCS, the anodal electrode placed over the left C2 nerve dermatome, and cathodal electrode placed over the right C2 dermatome. A constant current of 1.5 mA was applied for 20 min.
  Arms: Active ON-tDCS
Device: Sham ON-tDCS — For sham group, placement of the electrodes was identical to that of active ON-tDCS. ON-tDCS was first switched on in a ramp-up fashion over 5 s. Current intensity (ramp down) was gradually reduced (over 5 s) as soon as ON-tDCS reached a current flow of 1.5 mA. Hence, sham ON-tDCS only lasted 10 s (as opposed to 20 min in the active group).
  Arms: Sham ON-tDCS

SUMMARY:
So far, antidepressant drugs have limited memory improvement. Transcranial direct current stimulation, as a non-invasive and safe neuroregulatory technique, is a new direction to improve memory.In this study, transcranial direct current stimulation of the greater occipital nerve was used to explore the effect of improving memory function in patients with stable depression, and related studies were conducted on the locus coeruleus-noadrenal loop and the functional connection between locus coeruleus, hippocampus and amygdala.

DETAILED DESCRIPTION:
In this study, a randomized, controlled, double-blind design was adopted. Patients with depression were randomly divided into an intervention group and a control group to receive true or fake tDCS stimulation respectively. Clinical data, memory and other related cognitive function assessment, EEG, resting state fMRI, saliva and blood indicators were collected two weeks before and two weeks after the intervention, and followed up for eight weeks. Finally, data correlation analysis was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for ICD-10 depressive episode (F32) or recurrent depressive disorder (F33) diagnosis;
2. Antidepressant therapy for at least 8 weeks, with no antidepressant adjustment for nearly 2 months
3. HAMD-17 scores ≤ 7 points at the time of enrollment; CGI score ≦2;
4. Chief complaint of memory impairment, PDQ-D score of cognitive impairment ≧17 points;
5. Right-handed.

Exclusion Criteria:

1. A history of major physical diseases;
2. Have other mental disorders that meet the diagnostic criteria of ICD-10;
3. Hearing, color blindness, color weakness or receive electroconvulsive therapy;
4. Alcohol dependence or substance abuse;
5. Patients with intellectual disability;
6. Pregnant or lactating women or those planning to become pregnant;
7. Patients with contraindications to tDCS.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in working memory test scores after intervention. | Baseline, 2-week, 2-month
  The working memory test consists of two parts, which measure the breadth and accuracy of working memory respectively. The breadth of working memory will be tested using the operating span experiment, as the accuracy of working memory will be tested using the Memory Orientation experiment.

SECONDARY OUTCOMES:
Change in three component test of executive function scores after intervention. | Baseline, 2-week, 2-month
  The three component tests of executive function were one-backward test, anti-saccade and shifting test respectively.In the one-backward test, subjects need to memorize letters while counting numbers, scoring them according to the accuracy of the alphabetic memory order; The anti-saccade test asks subjects to react to a flash of arrows (0.5 seconds) by selecting the direction they see on a keyboard；The shifting test asked subjects to select a forward or reverse feedback key depending on where the icon appeared.
Change in the test of logical memory on the Wechsler Memory Test score after intervention. | Baseline, 2-week, 2-month
  The test asked participants to retell a story they had heard and rate how well they recalled it

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hanzhou, Zhejiang, China